CLINICAL TRIAL: NCT00659178
Title: A Phase I, Dose Escalation Study to Assess the Safety & Biological Activity of Interleukin 18 (SB-485232) Administered by IV Infusion in Combination With Pegylated Liposomal Doxorubicin (Doxil) in Advanced Stage Epithelial Ovarian Cancer
Brief Title: Combination Study Of SB-485232 (Interleukin 18) And Doxil For Advanced Stage Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILI108621
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms, Ovarian
Keywords: Doxil,; pegylated liposomal doxorubicin,; ovarian cancer; IL-18,; combination study,; immunotherapy,; cytokine,
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Interleukin-18; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB-485232 plus pegylated liposomal doxorubicin (Experimental): Subjects will receive one dose of pegylated liposomal doxorubicin on Day 1 plus two doses of SB-485232 on Day 3 and Day 9 in each cycle.
  Interventions: Drug: SB-485232 (interleukin 18), pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: SB-485232 (interleukin 18), pegylated liposomal doxorubicin — SB-485232 (interleukin 18), pegylated liposomal doxorubicin
  Other Names: SB-485232 (interleukin 18); pegylated liposomal doxorubicin

SUMMARY:
The purpose of this study is to identify a dose of SB-485232 which is safe, tolerable and biologically active when used in combination with pegylated liposomal doxorubicin (Doxil) in patients with epithelial ovarian cancer. This study will use a standard treatment regimen of pegylated liposomal doxorubicin (Doxil) in combination with rising doses of SB-485232. The dose selected from this study will be used in a future studies to evaluate the efficacy of this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age ≥18 years of age;
2. Histologically confirmed diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma;
3. Candidate to receive pegylated liposomal doxorubicin for treatment of advanced stage ovarian cancer as per standard of care and in the opinion of the treating principal investigator;
4. Measurable lesion(s) according to RECIST v1.0;
5. ECOG performance status of 0, 1 or 2;
6. Predicted life expectancy of ≥4 months
7. No chemotherapy, immunotherapy, hormonal therapy, or biological therapy for cancer, radiotherapy, or surgical procedures (except for minor surgical procedures) within four weeks before beginning treatment with SB-485232 (six weeks for nitrosoureas and mitomycin C). Subjects must have recovered from toxicities (incurred as a result of previous therapy) sufficiently to be entered into a Phase I study;
8. Disease-free period of at least five years from prior malignancies (except for curatively treated basal and squamous cell carcinomas of the skin and/or carcinoma of the cervix in situ);
9. Left ventricular ejection fraction (LVEF) ≥50 % as determined by MUGA scan;
10. A signed and dated written informed consent form is obtained from the subject;
11. The subject is able to understand and comply with protocol requirements, timetables, instructions and protocol-stated restrictions;
12. The subject is likely to maintain good venous blood access for PK and PD sampling throughout the study;
13. A female is eligible to enter and participate in the study if she is of: non-childbearing potential (i.e., physiologically incapable of becoming pregnant) or, childbearing potential, has a negative serum pregnancy test at the screening visit, and agrees to one of several GSK acceptable contraceptive methods;
14. Adequate organ function defined as: ANC ≥1.5 x 10^9/L; hemoglobin ≥9 g/dL (after transfusion if needed); platelets ≥75 x 10^9/L.

Exclusion Criteria:

1. Significant cardiac, pulmonary, metabolic, renal, hepatic, gastrointestinal or autoimmune conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as participant in this trial;
2. Any severe concurrent disease or condition, including significant active autoimmune diseases such as rheumatoid arthritis, which in the judgment of the principal investigator, would make the subject inappropriate for study participation;
3. History of myocardial infarction, unstable angina, or acute coronary syndrome within the past six months;
4. The subject has a history of hypersensitivity reactions to a conventional formulation of doxorubicin HCl or the components of pegylated liposomal doxorubicin;
5. The subject has a history of receiving a total cumulative dosage of doxorubicin HCl exceeding the currently recommended limit of 550 mg/m^2 or will exceed the 550 mg/m^2 dosage limit during the course of the current study. A subject will also be excluded if they received a lower cumulative dosage of doxorubicin HCl (i.e., 400 mg/m^2) and also had prior radiotherapy to the mediastinal area or concomitant therapy with other potentially cardiotoxic agents such as cyclophosphamide. Prior use of other anthracyclines or anthracenediones should be included in calculations of total cumulative doxorubicin HCl dosage;
6. Women who are pregnant or are breast-feeding;
7. Corrected QT interval (QTc) ≥480 msec (average of three measurements to be made at screening);
8. The subject has diabetes mellitus with poor glycemic control;
9. The subject has a history of human immunodeficiency virus (HIV) or other immunodeficiency disease;
10. The subject has positive Hepatitis B surface antigen;
11. The subject has a history of a severe infusion-related reaction following treatment with pegylated liposomal doxorubicin as described in the protocol;
12. The subject has an acute infection or severe or uncontrolled infections requiring systemic antibiotic therapy;
13. Any serious medical or psychiatric disorder that would interfere with subject safety or informed consent;
14. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol;
15. Known leptomeningeal disease or evidence of prior or current metastatic brain disease. Routine screening with central nervous system (CNS) imaging studies (CT or MRI) is required only if clinically indicated;
16. Receiving concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy;
17. Oral corticosteroids within 14 days of study entry;
18. History of ventricular arrhythmias requiring drug or device therapy;
19. Any investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of SB-485232;
20. The subject has active signs of a bowel obstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-06-18 (Actual); Primary Completion 2011-02-18 (Actual); Study Completion 2011-02-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SB-485232/Doxil combination therapy | 16 weeks

SECONDARY OUTCOMES:
Biological activity of SB-485232/Doxil combination therapy | 16 weeks
Pharmacokinetic parameters for SB-485232 and Doxil: AUC(0-t), Cmax, and Cmin | 16 weeks
Pharmacodynamic biomarker responses | 16 weeks
Immunogenicity (anti-SB-485232 and anti-PEG antibodies) | 16 weeks
Anti-tumor activity (Radiographic tumor assessments and serum CA-125 levels) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study ILI108621 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/ILI108621?search=study&search_terms=ILI108621#rs
- Available data/document: Statistical Analysis Plan: ILI108621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ILI108621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ILI108621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ILI108621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ILI108621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ILI108621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ILI108621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register